CLINICAL TRIAL: NCT03567811
Title: Exertional Exhaustion in Chronic Fatigue Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, James Baraniuk, MD, Professor of Medicine, Georgetown University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-0943
Record Dates: First submitted 2018-04-20; First posted 2018-06-26 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Intervention Model Description: All subjects were participated in an identical protocol. Outcomes were compared between control and Chronic Fatigue Syndrome subjects.
Masking Description: All control and Chronic Fatigue Syndrome subjects were treated in identical fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Fatigue Syndrome (Other): Inclusion and exclusion criteria based on 1994 Center for Disease Control ("Fukuda") criteria of persistent, disabling, moderate to severe fatigue that was relieved by rest, plus at least 4 of the 8 following ancillary features: cognitive dysfunction affecting short term memory or concentration, sore throat, sore lymph nodes, sore muscles, sore joints, headache, sleep disturbance, and exertional exhaustion (post-exertional malaise). Intervention: Procedure/Surgery: Submaximal bicycle exercise stress test on Days 1 and 2
  Interventions: Procedure: Submaximal bicycle exercise stress test on Days 1 and 2
- Sedentary Control (Other): Subjects who lived a sedentary lifestyle, did not meet Chronic Fatigue Syndrome criteria, and did not have any exclusionary chronic medical, psychiatric or other conditions were our Sedentary Control subjects. By design, this control group included controlled Type II diabetes and thyroid disease, chronic idiopathic fatigue, hypertension (other heart disease excluded) and other stable medical conditions. This variety of subjects were included to prevent ceiling (CFS) vs. floor (control) effects if the control group had totally pristine subjects with zero health issues. Intervention: Procedure/Surgery: Submaximal bicycle exercise stress test on Days 1 and 2
  Interventions: Procedure: Submaximal bicycle exercise stress test on Days 1 and 2

INTERVENTIONS:
Procedure: Submaximal bicycle exercise stress test on Days 1 and 2 — Identical submaximal stress tests were performed on both days to see if Day 1 exercise reduced performance on Day 2, or caused changes between BOLD scans during cognitive testing between Day 1 and Day 2.

SUMMARY:
Post-exertional malaise was modeled by having Chronic Fatigue Syndrome (CFS) and sedentary control subjects perform submaximal exercise on 2 consecutive days with objective changes in brain function measured by magnetic resonance imaging (MRI) during cognitive tests before and after the 2 exercise sessions.

DETAILED DESCRIPTION:
Chronic Fatigue Syndrome (CFS) and sedentary control subjects answered on-line advertisements and word-of-mouth communications. Candidates gave verbal informed consent to discuss their medical history during a telephone interview. If the met inclusion and exclusion criteria, they were assigned an log-in code and password to complete an extensive on-line questionnaire, and were scheduled for the 3 day in-patient study.

On the Screening Day subjects completed written informed consent, history and physical, screening blood work, mental status exam, heart rate variability for orthostasis, and dolorimetry for systemic hyperalgesia.

On Exercise Day 1, subjects had magnetic resonance imaging (MRI) for structure (MPRAGE), white matter integrity (diffusion tensor imaging, DTI), and blood oxygenation level dependent (BOLD) analysis during working memory tasks. The tasks were the simple stimulus-response 0-back "see a letter, push a button" task, and the difficult continuous 2-back task "see a string of letters, remember the letters in order, press the button for the letter seen 2 previously ("2-back)".

The submaximal exercise test was performed in identical fashion on day 1 and day 2. Subjects rested on a bicycle ergometer for 5 minutes for baseline cardiopulmonary (VO2) measurements. They began pedalling with resistance increased in step wise fashion until their heart rate reached 70% of predicted maximum heart rate (pHR = 220 - age). They pedaled 25 minutes at 70% or until they felt they had their personal maximum effort (e.g. Borg Exertional Scale 19/20). If they reached 25 minutes, then resistance was increased until they reached 85% of pHR. Continuous EKG, symptoms and VO2 were followed from rest until 5 minutes after peak exercise.

Heart rate variability and symptoms were assessed during recumbent and standing posture to assess orthostatic intolerance.

On Exercise Day 2, the same methods were used, but the order was reversed with the submaximal exercise test first, followed by the identical MRI protocol.

ELIGIBILITY:
Inclusion Criteria:

CFS and healthy subjects

Exclusion Criteria:

* HIV / AIDS subjects
* Pregnant women
* Lactation
* Cognitive impairment, mental retardation, severe head injury, stroke, proven multiple sclerosis, "melancholic" suicidal major depression, schizophrenia, Alzheimer's disease, "mild cognitive impairment" (MCI), other dementia, or other serious neurological diseases
* Brain injury. stroke, severe head injury (concussion, severe motor vehicle accidents), bleeding into brain, have been unconscious for more than 1 day (in a coma), seizures, brain inflammation such as multiple sclerosis or lupus.
* Metal implants such as prostheses, wires, plates, or screws that may heat up in the magnetic resonance imaging scanner and cause harm.
* Claustrophobia.
* Abnormal laboratory and questionnaire results.
* Heart, lung, kidney, arthritis, autoimmune, cancer, and other chronic illnesses, leg amputations heart attacks (myocardial infarction), coronary artery disease, abnormal heart rhythms, congestive heart failure, heart valve disease, uncontrolled high blood pressure or strokes, lung disease from smoking or other causes, painful, swollen or deformed joints related to arthritis or autoimmune diseases, weakness from nerve damage, kidney disease on dialysis, liver disease (alcoholic cirrhosis, hepatitis B, hepatitis C), inflammatory bowel disease (Crohn's disease, ulcerative colitis), or cancer Subjects may participate if they have well-controlled diabetes or thyroid disease.

Any other chronic disease with chronic pain, fatigue and thinking problems (cognitive impairment) that would limit the ability to complete the questionnaires and other tests.

* Amputation that would prevent bicycle exercise.
* Medications. Drugs that interfere with heart, lung, brain and nerve function
* Drinking and Smoking. You will have to stop caffeine (coffee, tea, soft drinks), alcohol, cannabis and nicotine products (smoking) for 3 days before the study, and the full period of the testing.
* Difficulties Drawing Blood.
* Children under the age of 18 years
* Incarcerated people (in jail)
* Alcohol or substance abuse in the past 6 months.
* English: Subjects must be able to speak and understand English to be able to understand the tests and other instructions during the study.
* Disruptive: Subjects who are disruptive or may reveal medical information about other subjects will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in blood oxygenation level dependent (BOLD) patterns of brain blood flow during cognitive testing | Day 1 (pre-exercise) and Day 2 (after 2nd exercise)
  MRI with cognitive tasks were performed before Day 1 exercise and compared to after the Day 2 exercise.

SECONDARY OUTCOMES:
Postural change in heart rate and heart rate variability after exercise | Before exercise. 1, 3, 8, 24 and 36 hours after exercise
  Heart rates were recorded while subjects resting supine for 5 minutes, and during 5 minutes of standing. The change in heart rate (deltaHR) was calculated.
Pressure-induced pain (systemic hyperalgesia) by dolorimetry | 10 am each day for 4 days
  A strain gauge (algometer, dolorimeter) was pressed over 18 traditional fibromyalgia tender point locations at a slow rate < kg/sec with the subject instructed to tell the operator to stop pushing as soon as they felt pain.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Katopol, Study Chair — IRB Director

IPD SHARING:
Plan to Share IPD: Yes
RedCap
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 2019
Access Criteria: open

REFERENCES:
- [Result] Garner R, Baraniuk JN. Orthostatic intolerance in chronic fatigue syndrome. J Transl Med. 2019 Jun 3;17(1):185. doi: 10.1186/s12967-019-1935-y. PMID 31159884
- [Result] Timbol CR, Baraniuk JN. Chronic fatigue syndrome in the emergency department. Open Access Emerg Med. 2019 Jan 11;11:15-28. doi: 10.2147/OAEM.S176843. eCollection 2019. PMID 30666170
- [Result] Rayhan RU, Ravindran MK, Baraniuk JN. Migraine in gulf war illness and chronic fatigue syndrome: prevalence, potential mechanisms, and evaluation. Front Physiol. 2013 Jul 24;4:181. doi: 10.3389/fphys.2013.00181. eCollection 2013. PMID 23898301
- [Result] Baraniuk JN. Chronic Fatigue Syndrome prevalence is grossly overestimated using Oxford criteria compared to Centers for Disease Control (Fukuda) criteria in a U.S. population study. Fatigue. 2017;5(4):215-230. doi: 10.1080/21641846.2017.1353578. Epub 2017 Jul 21. PMID 30854252
- [Result] Baraniuk JN, Shivapurkar N. Exercise - induced changes in cerebrospinal fluid miRNAs in Gulf War Illness, Chronic Fatigue Syndrome and sedentary control subjects. Sci Rep. 2017 Nov 10;7(1):15338. doi: 10.1038/s41598-017-15383-9. PMID 29127316
- [Result] Baraniuk JN, Shivapurkar N. Author Correction: Exercise - induced changes in cerebrospinal fluid miRNAs in Gulf War Illness, Chronic Fatigue Syndrome and sedentary control subjects. Sci Rep. 2018 Apr 19;8(1):6455. doi: 10.1038/s41598-018-23238-0. PMID 29674668